CLINICAL TRIAL: NCT01811368
Title: Use of Zevalin to Enhance the Efficacy of Non-Myeloablative Allogeneic Transplantation in Patients With Relapsed or Refractory CD20+ Non-Hodgkin's Lymphoma
Brief Title: Zevalin Before Stem Cell Transplant in Treating Patients With Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Joseph Tuscano (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 367905; UCDCC#233 (Other: UC Davis); NCI-2012-02753 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Refractory Non Hodgkin Lymphoma; Relapsed Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; ibritumomab tiuxetan; Antilymphocyte Serum; thymoglobulin; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibritumomab tiuxetan, allogeneic PBSCT) (Experimental): CONDITIONING REGIMEN: Patients receive rituximab IV on days -21 and 14, ibritumomab tiuxetan IV on day -14, TLI on days -11 to -7 and -4 to -1, and antithymocyte globulin IV over 4-6 hours on days -11 to -7. Patients also undergo TLI on days -11 to -7 and -4 to -1.
  TRANSPLANT: Patients undergo allogeneic PBSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclosporine PO BID or IV on days -3 to 56 with taper to 6 months and mycophenolate mofetil PO BID or IV on days 0-28.
  Interventions: Biological: rituximab; Biological: ibritumomab tiuxetan; Biological: anti-thymocyte globulin; Radiation: total nodal irradiation; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; Mabthera; Rituxan
Biological: ibritumomab tiuxetan — Given IV
  Other Names: Zevalin
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Radiation: total nodal irradiation — Undergo TLI
  Other Names: TLI; total lymphoid irradiation
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic peripheral blood stem cell transplant
Drug: cyclosporine — Given PO or IV
  Other Names: cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO or IV
  Other Names: Cellcept; MMF

SUMMARY:
This phase II trial studies how well ibritumomab tiuxetan before donor peripheral blood stem cell transplant works in treating patients with relapsed or refractory non-Hodgkin lymphoma. Giving rituximab, antithymocyte globulin, and total-lymphoid irradiation (TLI) before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. Also, radiolabeled monoclonal antibodies, such as ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving rituximab, antithymocyte globulin, and TLI before the transplant together with cyclosporine and mycophenolate mofetil after the transplant may stop this from happening. Giving a radiolabeled monoclonal antibody before a donor peripheral blood stem cell transplant may be an effective treatment for non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the response conversion (progressive disease [PD]/stable disease [SD] to partial response [PR] and complete response [CR]).

SECONDARY OBJECTIVES:

I. To assess the time to engraftment/chimerism. II. To assess the rate of acute and chronic graft-versus-host disease (GVHD). III. To assess toxicity. IV. To determine the overall survival. V. To investigate immune functional and phenotypic analysis. VI. To measure two year event free survival (EFS).

OUTLINE:

CONDITIONING REGIMEN: Patients receive rituximab intravenously (IV) on days -21 and 14, ibritumomab tiuxetan IV on day -14, TLI on days -11 to -7 and -4 to -1, and antithymocyte globulin IV over 4-6 hours on days -11 to -7. Patients also undergo TLI on days -11 to -7 and -4 to -1.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant (PBSCT) on day 0.

GVHD PROPHYLAXIS: Patients receive cyclosporine orally (PO) twice daily (BID) or IV on days -3 to 56 with taper to 6 months and mycophenolate mofetil PO BID or IV on days 0-28.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed relapsed cluster of differentiation (CD)20+ non-Hodgkin's lymphoma (NHL) (included in this category are follicular grade I, II, III, marginal zone, mantle cell, diffuse large B cell, small lymphocytic lymphoma) and CD20+ Hodgkin's disease for which standard curative therapy does not exist or is no longer effective
* Patients must have had at least one prior chemotherapeutic regimen; steroids alone and local radiation do not count as regimens; radiotherapy must have been completed at least 4 weeks prior to entry into the study; Rituxan alone does not count as a regimen; however, Bexxar or Zevalin (ibritumomab tiuxetan) do and patients must have completed radioimmunotherapy (RIT) > 12 months prior to enrollment
* Karnofsky performance status of ≥ 60%
* Life expectancy of greater than 3 months
* Total bilirubin within institutional normal limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Blood counts no restrictions
* Patients who had anything less than a CR (PR, SD or progressive disease) to their last salvage regimen
* Ability to understand and the willingness to sign a written informed consent document
* Patients fit for non-myeloablative transplantation or best treatment that have an available matched (9/10 or better) related or unrelated donor
* Patients who are considered rituximab refractory (defined as progression within 6 months of their last rituximab-containing regimen)

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, rituximab within three months (unless there is evidence of progression), or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are excluded; this does not include the use of steroids which may continue until two days prior to enrollment
* Patients may not be receiving any other investigational agents
* Failure to obtain insurance/payment authorization for Zevalin, unless the subject agrees to cover the cost
* Patients with known active brain metastases, other neurological disorders/dysfunction or a history of seizure disorder, or other neurological dysfunction should be excluded from this clinical trial because of their poor prognosis
* Patients who have an uncontrolled infection (presumed or documented) with progression after appropriate therapy for greater than one month
* Patients with symptomatic coronary artery disease, uncontrolled congestive heart failure; left ventricular ejection fraction is not required to be measured, however if it is measured, patient is excluded if ejection fraction is < 30%
* Patients requiring supplementary continuous oxygen; diffusion capacity of the lung of carbon monoxide (DLCO) is not required to be measured, however if it is measured, patient is excluded if DLCO < 35%
* Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function and histology, and for the degree of portal hypertension
* Patients with any of the following liver function abnormalities will be excluded:

  * Fulminant liver failure
  * Cirrhosis with evidence of portal hypertension or bridging fibrosis
  * Alcoholic hepatitis
  * Esophageal varices
  * A history of bleeding esophageal varices
  * Hepatic encephalopathy
  * Uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time
  * Ascites related to portal hypertension
  * Chronic viral hepatitis with total serum bilirubin > 3 mg/dL
  * Symptomatic biliary disease
* Pregnant women are excluded from this study
* Human immunodeficiency virus (HIV)-positive patients

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03-12 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Response conversion rate (PD/SD to PR and CR) | Up to 60 days post-transplant
  Calculated along with 95% confidence intervals (CI). Logistic regression will be used to assess the impact of patient characteristics (e.g., low/high lactate dehydrogenase isoenzyme-3 [LDH] or immunologic correlates) on the response conversion rate.

SECONDARY OUTCOMES:
Time to engraftment/chimerism | Up to 3 years
  Estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups of patients will be made using the logrank test. Cox (proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes when proper.
Rate of acute GVHD | Up to day 730
Rate of chronic GVHD | Up to day 730
Overall survival | Up to day 730
  Estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups of patients will be made using the logrank test. Cox (proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes when proper.
EFS | 2 years
  Comparison of time-to-event endpoints by important subgroups of patients will be made using the logrank test. Cox (proportional hazards) regression will be used to evaluate multivariable predictive models of time-to-event outcomes when proper.
Toxicities | Up to day 730
  Toxicities as measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tuscano, Principal Investigator — UC Davis Comprehensive Cancer Center
Locations (1):
- University of California Davis, Sacramento, California, United States